CLINICAL TRIAL: NCT05489640
Title: A Real-World Study to Determine Patient Characteristics, Treatment Patterns, Clinical and Patient-Reported Outcomes of Patients With Hereditary Angioedema That Self-Administered Icatibant Using Homecare Services in the UK
Brief Title: A Study in Adults With Hereditary Angioedema (HAE) Who Currently Receive Icatibant at Home
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-667-4002; MACS-2021-061502 (Other: Takeda)
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: Drug Therapy
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HAE Participants: Adult participants with a diagnosis of HAE who are receiving treatment according to routine clinical practice and prescribed all treatments in accordance with the approved marketing authorization will be enrolled in this study. Data will be directly collected from participants via patient reported diaries and paper- based and/or electronic homecare records as appropriate for UK participants using homecare services for icatibant. No study specific intervention will be administered in this study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention will be administered in this study.

SUMMARY:
The main aim of this study is to describe the treatment patterns, characteristics and outcomes of people with HAE who are currently receiving icatibant in the homecare setting in the United Kingdom (UK).

Participants will be treated with icatibant according to their routine practice via homecare service for icatibant within the UK. Data will be directly collected from participants via study diaries and questionnaires. Participants will be contacted approximately every 90 days during study duration (this can occur via phone or as a face-to-face visit).

ELIGIBILITY:
Inclusion Criteria

* Participants self-administering or receiving care assisted administration of icatibant treatment for patient confirmed diagnosis of HAE Type I or II in the homecare setting
* Participants who are able and willing to complete the study questionnaires
* Participants who are willing to be visited or contacted by a member of the homecare or research team at pre-arranged intervals in order to complete questionnaires

Exclusion Criteria

- Participants who have received icatibant as an investigational medicine as part of a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with a diagnosis of HAE I or II who are receiving treatment according to routine clinical practice and prescribed all treatments in accordance with the approved marketing authorization will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants Treated with Icatibant in the Homecare Setting who Were Receiving Prophylaxis Treatment at Index | Up to 12 months from Index (day of the first homecare telephonic consultation/visit)
Number of Participants Treated with Icatibant in the Homecare Setting in Each Prophylactic Treatment Type | Up to 12 months from Index (day of the first homecare telephonic consultation/visit)

SECONDARY OUTCOMES:
Number of Participants Categorized by Their Demographic Characteristics | Baseline Period [3 months prior to Index (day of the first homecare telephonic consultation/visit)]
  Demographic characteristics will include age at index (categories: 18-29, 30-39, 40-49, 50-59, 60+ years), sex (male, female, non-binary), and ethnic group.
Number of Participants Categorized by Their Clinical Characteristics | At Index (day of the first homecare telephonic consultation/visit)
  Clinical characteristics will include patient reported HAE type (Type I or Type II), categories of duration (participant's self-administration of icatibant at home and time since HAE diagnosis) at index, comorbidities, prior HAE related concomitant medication details, categories of details of deaths during the study observation period.
Rate of New HAE Attacks | Up to 12 months from Index (day of the first homecare telephonic consultation/visit)
  Rate of new HAE attacks and rate of new HAE attacks that required treatment in homecare setting will be recorded as number of HAE attacks per participant per month. Data would be reported for pre-defined time-period categories as follows:
  between index to month 3, between month 3 to 6, month 6 to 9 and month 9 to 12.
Frequency of Visits to Accident and Emergency Services Related to an HAE Attack | Up to 12 months from Index (day of the first homecare telephonic consultation/visit)
  Frequency of visits to Accident and Emergency Services related to an HAE attack will be defined as number of visits to Accidents and Emergency Services during pre-defined time period. Data would be reported for pre-defined time-period categories as follows: between index to month 3, between month 3 to 6, month 6 to 9 and month 9 to 12.
Time from the Start of Each HAE Attack to Administration of Icatibant in the Homecare Setting | Up to 12 months from Index (day of the first homecare telephonic consultation/visit)
  The summary data for time (in hours) from the start of each HAE attack to administration of icatibant in the homecare setting will be reported.
Frequency of Icatibant Administration Following Start of Each HAE Attack | Up to 12 months from Index (day of the first homecare telephonic consultation/visit)
  The summary data for number of icatibant administration following start of each HAE attack during the predefined time period will be reported.
Number of Participants by Treatment Patterns | Up to 12 months from Index (day of the first homecare telephonic consultation/visit)
  Treatment patterns will include assessment of number of participants by treatment dose received for HAE attack and average dose per participant received post-index.
Number of Participants by Treatment Management Patterns | Up to 12 months from Index (day of the first homecare telephonic consultation/visit)
  Treatment management patterns will include assessment of number of participants by discontinuations of icatibant treatment and reasons for discontinuation (this would be assessed for participants who received prophylaxis treatment during the study), number of face-to-face and telephone-based homecare consultations.
EQ-5D-5L Score | Up to 12 months from Index (day of the first homecare telephonic consultation/visit)
  The EQ-5D-5L questionnaire will be used to record impact of HAE on participant's quality-of-life (QoL). The EQ-5D-5L is a descriptive system of Health-Related Quality-of-Life (HRQoL) states consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each of which can take 1 of 5 responses. The responses record 5 levels of severity [no problems, slight problems, moderate problems, severe problems, and extreme problems] within a particular dimension. The scores will be the sum of scores from each dimension and can range from 5 (no problems) to 25 (extreme problems).
AE-QoL Total Score | Up to 12 months from Index (day of the first homecare telephonic consultation/visit)
  The Angioedema Quality of Life (AE-QoL) includes 17 items and 4 domains: functioning, fatigue/mood, fears/shame, and food. Raw scores from each domain will be linearly transformed to a total score of 0 to 100, with higher scores indicating a stronger impairment.
Angioedema Control Test (AECT) Total Score | Up to 12 months from Index (day of the first homecare telephonic consultation/visit)
  The AECT is used to assess participants with recurrent angioedema. The test uses a questionnaire with 4 items, each of which has 5 options and is used to measure the participant's current disease control. HAE control score will be recorded with 5 levels of answers [1=very often, 2=often, 3=sometimes, 4=seldom, 5=not at all] to the following questions: 1) In the last 3 months, how often have you had angioedema? 2) In the last 3 months, how much has your QoL been affected by angioedema? 3) In the last 3 months, how much has the unpredictability of your angioedema bothered you? 4) In the last 3 months, how well has your angioedema been controlled by your therapy? The total scores are the sum of individual scores from 4 items and will range from 4 (Very often) to 20 (not at all). Higher scores will indicate no recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Sciensus, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/ba1ce272a46640c4?idFilter=%5B%22TAK-667-4002%22%5D